CLINICAL TRIAL: NCT00905905
Title: Additive Effect of Ezetimibe Upon Simvastatin Treatment on Systemic Inflammatory Activity and Endothelial Function During Myocardial Infarction
Brief Title: Additive Effect of Ezetimibe Upon Simvastatin During Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia Heart Study Group (Other)
Responsible Party: Andrei C. Sposito, University of Brasilia Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EMI
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; systemic inflammatory activity; endothelial function
MeSH Terms: conditions — Myocardial Infarction | interventions — Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe-Simvastatin 10/40 mg (Experimental)
  Interventions: Drug: Ezetimibe-Simvastatin
- Simvastatin 40 mg (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40 mg/day during the first 7 days and then 20 mg/day for 3 more weeks until the evaluation of flow-mediated brachial artery dilation
  Other Names: Statin; Zocor
  Arms: Simvastatin 40 mg
Drug: Ezetimibe-Simvastatin — Ezetimibe-Simvastatin 10-40 mg/day during the first 7 days and then 20 mg/day for 3 more weeks until the evaluation of flow-mediated brachial artery dilation
  Other Names: Vytorin
  Arms: Ezetimibe-Simvastatin 10/40 mg

SUMMARY:
During acute coronary syndromes (ACS), the generation of inflammatory mediators negatively influences arterial wall remodeling and the endothelium-dependent vasomotor function in the coronary and systemic arterial systems. In fact, the intensity of the inflammatory upregulation is strongly related to the incidence of recurrent coronary events. The investigators previously demonstrated that high dose potent statins can rapidly reduce plasma levels of cholesterol-rich lipoproteins and inflammatory activity in subjects during ACS. In addition, such statin treatment attenuates the post-discharge endothelial dysfunction of these patients. By inference, it is plausible to hypothesize that these beneficial effects during ACS may be intensified by an additive lowering of plasma cholesterol through the treatment with ezetimibe. So far, data is unavailable to verify this assumption. In parallel, data from animal models have suggested that both statins and ezetimibe may reduce insulin sensitivity by their effect on cholesterol content and, by this way, on insulin signaling in liver cells. In this context, the present study aims to investigate the role of the addition of ezetimibe upon statin treatment on stress-induced insulin resistance and on the time-course of the inflammatory response during the acute phase of myocardial infarction and its late effect on endothelium-dependent arterial dilation.

ELIGIBILITY:
Inclusion Criteria:

* less than 24 hours after the onset of myocardial infarction symptoms
* ST-segment elevation of a least 1 mm (frontal plane) or 2 mm (horizontal plane) in two contiguous leads
* myocardial necrosis, as evidenced by increased CK-MB and troponin levels

Exclusion Criteria:

* use of statins for the last 6 months before myocardial infarction

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
C- reactive Protein (CRP) elevation during the first 7 days after myocardial infarction | 5th day

SECONDARY OUTCOMES:
Endothelial function 30 days after myocardial infarction | 30th day
Stress Insulin Resistance | 5th day
  Evaluation of the change in plasma glucose, insulin and C-peptide from admission to the fifth day after myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, MD, PhD, Study Chair — University of Brasilia Medical School
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil